CLINICAL TRIAL: NCT03753139
Title: Identification of Arrhythmias With One-time ECG
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Other Study IDs: KUH507P002
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation; Heart Rate Fast; Heart Rate Low
Keywords: Atrial fibrillation; detection; portable device; algorithms
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia; Bradycardia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial fibrillation: Patients with atrial fibrillation as recorded by Holter
  Interventions: Device: Heart rhythm monitoring with portable device
- Sinus rhythm: Patients with sinus rhythm as recorded by Holter
  Interventions: Device: Heart rhythm monitoring with portable device

INTERVENTIONS:
Device: Heart rhythm monitoring with portable device — The study compares the ability of lightweight measurement methods to detect different heart rhythms compared to the Holter registration.
  1. Faros 360 ECG sensor with wet electrodes. Faros 360 Holter is CE and FDA 510 cleared class 2a medical device, which is attached to the patient's chest with five single-use wet electrodes.
  2. Suunto Movesense one-time ECG device (Suunto Oy, http://www.suunto.com Vantaa Finland). Movesense is CE cleared consumer device, which is used with two dry electrodes to the ECG measurement.
  3. Empatica E4 activity bracelet (Empatica Ltd http://www.empatica.com Milan, Italy), which is CE cleared consumer device. Empatica E4 is a photopletysmogram which measures optically the amount of blood circulating in the blood vessel.
  4. Samsung Gear S3 wearable (Samsung Electronics, Co., Soul, South Korea) which is CE cleared consumer device. Gear S3 is a photopletysmogram, which measures optically the amount of blood circulating in the blood vessel.

SUMMARY:
In Western countries, every sixth person in their lifetime and 15,000 people in Finland have a new stroke each year. About every fourth stroke is based on cardiac embolism. Atrial fibrillation causes formation of thrombi in the left atrium with ensuing embolization in the cerebral and peripheral circulation.

This study investigates the suitability of measurement techniques and new calculation methods used in sport/wellness technology for the screening and diagnosis of atrial fibrillation and other arrhythmias. New measurement technologies, the one-time ECG measurement and pulse wristband measurement, are studied for their characteristics, data quality and rhythm recognition. Identifying latent arrhythmias with new self-monitoring technologies can significantly reduce the number of strokes (the latent arrhythmias causes about 25% of strokes).

The research will be accomplished in cooperation with the Kuopio University Hospital Emergency Department, the Heart Center, the Department of Applied Physics of the University of Eastern Finland and Heart2Save Ltd.

The results of the research project will be published in the scientific journals of medicine and medical technology and will be presented at scientific conferences of the respective fields. The research results of the project can be utilized by all companies in the medical technology industry, in particular companies that produce ECG measuring instruments and companies that produce rhythm recognition software.

DETAILED DESCRIPTION:
The research aims to solve the following medical problems:

1. Identifying and defining the type of atrial fibrillation is problematic due to its spontaneous occurrence and latency.
2. Measurement devices for screening atrial fibrillation are poorly available.

The main research questions are:

1. Can a single-lead ECG measurement be used to detect arrhythmias

   1. Find out the measurement locations (ECG leads) for single-lead ECG self-monitoring and evaluate the impact of measurement locations on usability and signal quality.
   2. Find out the measurement locations for single-lead ECG monitoring when the measurement is performed by another person (nurse or relative) and evaluate the impact of measurement locations on usability and signal quality.
   3. Find out the reliability of single-lead ECG measurement for the identification of atrial fibrillation.
   4. Find out the reliability of single-lead ECG measurement for identification of rapid (tachycardia) and slow heart rate (bradycardia).
2. Can a wristband based on optical pulse registration be able to obtain reliable information about arrhythmias

   1. Find out the usability of the pulse wristband for the identification of atrial fibrillation.
   2. Find out the usability of the pulse wristband for the identification of rapid (tachycardia) and slow heart rate (bradycardia).

The purpose of the study's method development is to evaluate reliability of heart rate measurement in single-lead ECG and pulse wave measurement with healthy and patients with heart problems. The study develops computing methods based on lightweight measurement technology to reliably identify the most common cardiac arrhythmia, atrial fibrillation. The diagnosis and treatment of atrial fibrillation are decisive factors for preventing strokes.

Research patients have already undergone a 12-channel clinical ECG registration included in the normal treatment process. This 12-channel ECG is used for the identification of patients suitable for research and dividing to subgroups (normal rhythm, atrial fibrillation, rapid or slow rhythm).

In actual study measurements, a Holter-ECG device is attached on patient's chest using five wet electrodes to be used as golden standard for rhythm monitoring. The lightweight measurement methods are compared with the result of the Holter-ECG registration. In addition, photopletysmogram is placed on patient's wrist for PPG registration. Figure 1 shows illustrative examples of the study's measurements.

The researcher measures one minute recordings from two different measuring positions (flank and chest) with a one-time ECG measuring device. After that, the patient performs one minute self-monitoring measurements with one-time ECG device from the all three positions (thumbs, flank and chest) and also from the chest with jewel-ECG.

The study compares the ability of these lightweight measurement methods to detect different heart rhythms compared to the Holter registration.

The devices used for the measurement are:

1. Faros 360 EKG sensor with wet electrodes (figure 1, device 1) (Mega Elektroniikka, http://www.megaemg.com/ Kuopio Suomi). Faros 360 Holter is CE and FDA 510(k) cleared class 2a medical device, which is attached to the patient's chest with five single-use wet electrodes.
2. Suunto Movesense one-time ECG device (Suunto Oy, http://www.suunto.com Vantaa Suomi). Movesense is CE cleared consumer device, which is used with two dy electrodes to the ECG measurement (Figure 1 devices 2 and 3). Movesense case; jewel and one-time ECG case.

   1. In the previous study (Afib24h), Valvira was reported and the research received permission for the clinical device study (Movesense + chest strap combination).
   2. For this study, Valira is reported for a clinical device study (Movesense + one-time ECG device combination)
3. Empatica E4 activity bracelet (Empatica Ltd http://www.empatica.com Milan Italia), which is CE cleared consumer device. Empatica E4 is also a photopletysmogram, which measures optically the amount of blood circulating in the blood vessel (Figure 1 device 4).
4. Samsung Gear S3 wearable (Samsung Electronics, Co., Ltd., www.samsung.com Soul Etelä-Korea) which is CE cleared consumer device. Gear S3 is also a photopletysmogram, which measures optically the amount of blood circulating in the blood vessel.

The researcher attaches devices to the patient. After that, the researcher starts a 10-minute registration with Faros 360 (device 1) and Empatica E4 (device 4) devices. During a 10-minute measurement, the researcher measures one minute recordings from two different measuring positions with the Movesense ECG (device 2) 1. from the chest, sternum perpendicularly 2. from the chest, along the sternum. The patient then carries out one minute self-monitoring measurements 1. from the chest, sternum perpendicularly 2. from the chest, along the sternum 3. from the lower part of the flank 4. from thumbs and 5. from the chest with a jewel-ECG.

Heart rate detection by ECG measurement is most commonly done by the detection of QRS complexes. Numerous of these QRS detectors have been developed in recent decades. ECG measurement with dry electrodes involves considerably more movement disturbances, compared to the wet electrode measurements, as even the small movements of the device induce major changes to the ECG signal. In addition, especially when using thumbs as a measurement points, the EMG noise from the muscles is remarkably high compared to the wet electrode measurements.

This project utilizes the methods developed in the earlier mobile-ECG-project for noise and QRS detection to allow reliably detection of QRS complexes and heart rate irregularities in the dry electrode measurements.

In this study, the previously developed heart rate detection methods are validated by study's measurements of normal sinus rhythm, atrial fibrillation, and slow (bradycardia) and rapid (tachycardia) heart rate.

This study examines capability of pulse detection in detection of atrial fibrillation. The photopletysmogram measures the absorption of light in the tissue. The absorption of light into the blood is greater than the absorption into the surrounding tissue. When the heart beats, capillaries expand and contract based on blood volume changes. Photopletysmography allows the heart rate measurement by detecting changes in absorption.

Photopletysmgram, like a mobile-ECG device, is particularly sensitive to motion, even the small motion of led/photodiode induce major change in light intensity.

Also, physiological changes cause a disturbance in heart rate measurement, for example, as the vascular elasticity changes, the pulse time changes, resulting a disturbance in measurement.

Unlike the high-frequency pierced QRS complex, the pulse wave is a low-frequency up-down variation, which causes its own challenges for accurate heart rate measurement.

The atriums work insufficiently in atrial fibrillation therefore the ventricles are not completely filled with blood. In addition, atrial fibrillation causes the irregular conduction of impulses from atriums to the ventricles leading to pulse irregularity. The amount of blood pumped varies from one stroke to stroke, which makes the pulse wave detection challenging.

This project develops methods for accurate heart rate measurement from a pulse wave series.

The method development aims to take account of disturbances due to the motion of the meter, pulse wave irregularities typical of atrial fibrillation, and the challenges of slow (bradycardia) and rapid (tachycardia) heart rate detection.

The main goal of the method development is to determine the pulse so precisely that pulse irregularity due to atrial fibrillation can be distinguished from normal sinus rhythm and reliably detect rapid and slow heart rhythms.

In atrial fibrillation, electrical impulses conduct randomly to the ventricles, causing the heart rate to be irregular and uneven. A large campaign by the Heart Association "Feel your pulse - prevent the stroke" is based on heart rate or pulse recognition. Pulse recognition is of course the cheapest method to detect atrial fibrillation, but this method produces a large number of false positives. By ECG measurement, the detection of atrial fibrillation is much more reliable. Automated atrial fibrillation detection algorithms have been developed for this purpose.

Identification of the atrium activation in long-term Holter-ECG measurements is generally very challenging due to the poor signal-noise-ratio (motion, muscle-artefacts and partly overlapping much stronger ventricular activity). For this reason, most atrial fibrillation detection algorithms are based on the identification of pulse irregularity. For parametrization of the irregularity of the heart rate (RR-interval) has been introduced several relatively simple but reliable time-level methods. As an example, A RdR-based method wherein the RR intervals (heart rate) are represented as a function of consecutive RR interval changes (heart rate change) (Lian et al. 2011). The RdR-graph defines the fragmentation of the pattern resulting from irregular heart rate changes. In addition, there are methods that estimate RR time series internal coherence (Lee et al. 2011). Various nonlinear methods have also been introduced to parametrization of the heart rate variation, enabling the dynamics of the heart rate variation to be described more broadly (without limitation of the linearity assumption). One class of nonlinear methods are different entropy quantities, these are particularly interesting for the identification of atrial fibrillation and the irregular heart rate. Entropy quantities can be used to estimate the regularity and predictability of the RR time series. Typically, the reliable calculation of the entropy quantities requires a relatively long measurement time, but also entropy quantities that are suitable for the analysis of short measurements have been introduced (Lake & Moorman 2011).

This research project develops new atrial fibrillation detection algorithms for the mobile-ECG measurement and pulse wave measurement on the basis of already existing methods. Algorithms must take into account atrial and ventricular premature complexes. Ignoring of these increases the irregularity of the RR time series and thus increases the number of false positive atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for any reason in the emergency department of Kuopio University Hospital.

Exclusion Criteria:

* body mass index (BMI) over 35, implanted heart pacemaker device and a medical condition requiring immediate treatment that would be delayed by the study measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 patients will be recruited in the research: 100 patients with normal sinus rhythm, 100 with atrial fibrillation, 50 with rapid rhythm (tachycardia, resting heart rate > 100 bpm) and 50 slow rhythms (bradycardia, resting heart rate< 50bpm).
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Heart rhythm monitoring with single-lead ECG | 30 minutes
  Sensitivity and Specificity for the atrial fibrillation detection

CONTACTS AND LOCATIONS:
Overall Officials: Tero J Martikainen, MD. PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio university hospital, Kuopio, Eastern-Finland, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amann A, Tratnig R, Unterkofler K. Reliability of old and new ventricular fibrillation detection algorithms for automated external defibrillators. Biomed Eng Online. 2005 Oct 27;4:60. doi: 10.1186/1475-925X-4-60. PMID 16253134
- [Background] Barro S, Ruiz R, Cabello D, Mira J. Algorithmic sequential decision-making in the frequency domain for life threatening ventricular arrhythmias and imitative artefacts: a diagnostic system. J Biomed Eng. 1989 Jul;11(4):320-8. doi: 10.1016/0141-5425(89)90067-8. PMID 2755113
- [Background] Cabello D, Barro S, Salceda JM, Ruiz R, Mira J. Fuzzy K-nearest neighbor classifiers for ventricular arrhythmia detection. Int J Biomed Comput. 1991 Feb;27(2):77-93. doi: 10.1016/0020-7101(91)90089-w. PMID 2032755
- [Background] Chen SW. A two-stage discrimination of cardiac arrhythmias using a total least squares-based prony modeling algorithm. IEEE Trans Biomed Eng. 2000 Oct;47(10):1317-27. doi: 10.1109/10.871404. PMID 11059166
- [Background] al-Fahoum AS, Howitt I. Combined wavelet transformation and radial basis neural networks for classifying life-threatening cardiac arrhythmias. Med Biol Eng Comput. 1999 Sep;37(5):566-73. doi: 10.1007/BF02513350. PMID 10723893
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S; Task Force on Practice Guidelines, American College of Cardiology/American Heart Association; Committee for Practice Guidelines, European Society of Cardiology; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation-executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients with Atrial Fibrillation). Eur Heart J. 2006 Aug;27(16):1979-2030. doi: 10.1093/eurheartj/ehl176. No abstract available. PMID 16885201
- [Background] Ge D, Srinivasan N, Krishnan SM. Cardiac arrhythmia classification using autoregressive modeling. Biomed Eng Online. 2002 Nov 13;1:5. doi: 10.1186/1475-925x-1-5. PMID 12473180
- [Background] Jekova I. Comparison of five algorithms for the detection of ventricular fibrillation from the surface ECG. Physiol Meas. 2000 Nov;21(4):429-39. doi: 10.1088/0967-3334/21/4/301. PMID 11110242
- [Background] Lake DE, Moorman JR. Accurate estimation of entropy in very short physiological time series: the problem of atrial fibrillation detection in implanted ventricular devices. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H319-25. doi: 10.1152/ajpheart.00561.2010. Epub 2010 Oct 29. PMID 21037227
- [Background] Lee J, Nam Y, McManus DD, Chon KH. Time-varying coherence function for atrial fibrillation detection. IEEE Trans Biomed Eng. 2013 Oct;60(10):2783-93. doi: 10.1109/TBME.2013.2264721. Epub 2013 May 22. PMID 23708769
- [Background] Li C, Zheng C, Tai C. Detection of ECG characteristic points using wavelet transforms. IEEE Trans Biomed Eng. 1995 Jan;42(1):21-8. doi: 10.1109/10.362922. PMID 7851927
- [Background] Lian J, Wang L, Muessig D. A simple method to detect atrial fibrillation using RR intervals. Am J Cardiol. 2011 May 15;107(10):1494-7. doi: 10.1016/j.amjcard.2011.01.028. Epub 2011 Mar 17. PMID 21420064
- [Background] Lipponen JA, Tarvainen MP, Laitinen T, Lyyra-Laitinen T, Karjalainen PA. A principal component regression approach for estimation of ventricular repolarization characteristics. IEEE Trans Biomed Eng. 2010 May;57(5):1062-9. doi: 10.1109/TBME.2009.2037492. Epub 2010 Feb 5. PMID 20142157
- [Background] Lipponen JA, Kemppainen J, Karjalainen PA, Laitinen T, Mikola H, Karki T, Tarvainen MP. Dynamic estimation of cardiac repolarization characteristics during hypoglycemia in healthy and diabetic subjects. Physiol Meas. 2011 Jun;32(6):649-60. doi: 10.1088/0967-3334/32/6/003. Epub 2011 Apr 20. PMID 21508439
- [Background] Lipponen JA, Tarvainen MP. Principal component model for maternal ECG extraction in fetal QRS detection. Physiol Meas. 2014 Aug;35(8):1637-48. doi: 10.1088/0967-3334/35/8/1637. Epub 2014 Jul 29. PMID 25069651
- [Background] Meretoja A, Roine RO, Kaste M, Linna M, Juntunen M, Erila T, Hillbom M, Marttila R, Rissanen A, Sivenius J, Hakkinen U. Stroke monitoring on a national level: PERFECT Stroke, a comprehensive, registry-linkage stroke database in Finland. Stroke. 2010 Oct;41(10):2239-46. doi: 10.1161/STROKEAHA.110.595173. Epub 2010 Aug 26. PMID 20798363
- [Background] Syvaoja S, Castren M, Mantyla P, Rissanen TT, Kivela A, Uusaro A, Jantti H. The feasibility of recognizing the heart rhythm with an automated external defibrillator from an area the size of a mobile phone. Eur J Emerg Med. 2016 Apr;23(2):102-7. doi: 10.1097/MEJ.0000000000000214. PMID 25325408
- [Background] Tarvainen MP, Ranta-Aho PO, Karjalainen PA. An advanced detrending method with application to HRV analysis. IEEE Trans Biomed Eng. 2002 Feb;49(2):172-5. doi: 10.1109/10.979357. PMID 12066885
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Thakor NV, Zhu YS, Pan KY. Ventricular tachycardia and fibrillation detection by a sequential hypothesis testing algorithm. IEEE Trans Biomed Eng. 1990 Sep;37(9):837-43. doi: 10.1109/10.58594. PMID 2227970
- [Background] Zhang XS, Zhu YS, Thakor NV, Wang ZZ. Detecting ventricular tachycardia and fibrillation by complexity measure. IEEE Trans Biomed Eng. 1999 May;46(5):548-55. doi: 10.1109/10.759055. PMID 10230133
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Alexandru Popescu B, Schotten U, Van Putte B, Vardas P. 2016 ESC Guidelines for the Management of Atrial Fibrillation Developed in Collaboration With EACTS. Rev Esp Cardiol (Engl Ed). 2017 Jan;70(1):50. doi: 10.1016/j.rec.2016.11.033. No abstract available. English, Spanish. PMID 28038729
- [Derived] Valiaho ES, Kuoppa P, Lipponen JA, Hartikainen JEK, Jantti H, Rissanen TT, Kolk I, Pohjantahti-Maaroos H, Castren M, Halonen J, Tarvainen MP, Santala OE, Martikainen TJ. Wrist Band Photoplethysmography Autocorrelation Analysis Enables Detection of Atrial Fibrillation Without Pulse Detection. Front Physiol. 2021 May 7;12:654555. doi: 10.3389/fphys.2021.654555. eCollection 2021. PMID 34025448
- [Derived] Santala OE, Lipponen JA, Jantti H, Rissanen TT, Halonen J, Kolk I, Pohjantahti-Maaroos H, Tarvainen MP, Valiaho ES, Hartikainen J, Martikainen T. Necklace-embedded electrocardiogram for the detection and diagnosis of atrial fibrillation. Clin Cardiol. 2021 May;44(5):620-626. doi: 10.1002/clc.23580. Epub 2021 Feb 25. PMID 33629410